CLINICAL TRIAL: NCT00716508
Title: Surgical Treatment for Acute Patella Tendon Rupture: a Prospective, Randomized Study Comparing Transpatellar Suture Tunnels Method vs. Suture Anchors.
Brief Title: Surgical Treatment for Acute Patella Tendon Rupture
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Our PI left our institutions as we could not longer continue.
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Kyle Webb, Research Administrator, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00010200
Record Dates: First submitted 2008-07-15; First posted 2008-07-16 (Estimated); Last update posted 2013-09-19 (Estimated); Status verified 2013-09

CONDITIONS: Acute Patella Tendon Rupture
Keywords: Patella tendon rupute, suture anchors, repair patella tendon
MeSH Terms: interventions — Wound Healing; Suture Anchors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Repair with suture anchors: The insertion points for the three suture anchors will be marked with electrocautery. The anchors will be placed approximately 2 mm from the articulate surface; placing them too superficially may increased the joint reactive force and lead to abnormal patella femora joint mechanics. Pilot holes will be drilled with a 3.2-mm drill bit parallel to the patella, avoiding penetration of the articular surface. Three Suture anchors (Arthrex, Naples FL) will be threaded with two No. 5 Fiberwire (Arthrex, Naples FL) sutures and will be inserted and deployed in the pilot holes in the usual manner.
  Interventions: Procedure: Repair with suture anchors.
- B (Active Comparator): Repair with transpatellar tunnels: We will make a small horizontal trough at the inferior pole of the patella. Multiple, braided Krackow sutures will then be placed through the substance of the tendon using no. 5 Fiberwire (Arthrex, Naples FL) suture. Three to four drill holes will then be made through the patella. Using a suture passer, the sutures will then be brought from distal to proximal and tied over the superior pole. The knee will be flexed to 45 degrees. The tendon will be repaired adjacent to the articular surface and not to the anterior surface of the patella.
  Interventions: Procedure: Repair with transpatellar tunnels

INTERVENTIONS:
Procedure: Repair with transpatellar tunnels — Repair with transpatellar tunnels: We will make a small horizontal trough at the inferior pole of the patella. Multiple, braided Krackow sutures will then be placed through the substance of the tendon using no. 5 Fiberwire (Arthrex, Naples FL) suture. Three to four drill holes will then be made through the patella. Using a suture passer, the sutures will then be brought from distal to proximal and tied over the superior pole. The knee will be flexed to 45 degrees. The tendon will be repaired adjacent to the articular surface and not to the anterior surface of the patella.
  Arms: B
Procedure: Repair with suture anchors. — Repair with suture anchors: The insertion points for the three suture anchors will be marked with electrocautery. The anchors will be placed approximately 2 mm from the articulate surface; placing them too superficially may increased the joint reactive force and lead to abnormal patella femora joint mechanics. Pilot holes will be drilled with a 3.2-mm drill bit parallel to the patella, avoiding penetration of the articular surface. Three Suture anchors (Arthrex, Naples FL) will be threaded with two No. 5 Fiberwire (Arthrex, Naples FL) sutures and will be inserted and deployed in the pilot holes in the usual manner.
  Arms: A

SUMMARY:
We will compare two groups for acute patella tendon repair: one treated with surgical anchors and the second, with transpatellar tunnels.

DETAILED DESCRIPTION:
The patella tendon is located in the knee, and is attached to the leg bone and the patella bone (knee cap). The quadriceps muscle (an important tight muscle) attaches to the patella bone and allows for extension and flexion of the leg. Rupture of the patella tendon occurs mainly in people under the age of 40 years old with an active lifestyle. Normally, surgical repair is needed to fix this injury. The widely accepted surgery for this injury consists in drilling 2 holes in the patella bone that are used to anchor the patella tendon in place. This surgery has some complications such as re-rupture of the tendon, breakage of the bone, etc. Some investigators have tried different techniques to avoid these complications with variable results. We want to use 2 anchors in the bone to avoid making holes in the patella bone, decreasing complications and surgical time, and hopefully, allowing for a better surgical repair. We will have 2 arms. One group will have the standard of care technique and the second group will have the anchors technique. We will follow up with our patients after the surgery to record their progress, and complications, if any. We will also have a standardized physical therapy program for consistency and to avoid any problems.

ELIGIBILITY:
Inclusion Criteria:

1. Stage of Disease: Acute ruptures of the patella tendon, no more than 3 weeks since the time of injury.
2. Age: 18 years old and up.
3. Performance status: Patients with no other previous illnesses that prevented them to ambulate normally (without help of devices).
4. Informed consent requirements: One person from our research staff will approach the patient after the diagnosis has been made. The diagnosis will be made by the doctor in charge on the patient care based on the medical history, physical exam and image studies (MRI). We will explain the benefits/risks to be part of the study and that they are not obligated to be part of it as part of their care.

Exclusion Criteria:

1. Prior treatment: Patients with chronic patella tendon ruptures (more than 3 weeks).
2. Prior other diseases: diseases with systemic collagen deficiencies.
3. Infection: Patients with active infection will be disqualified.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2008-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Outcome measures will include SF 36, Tegner and Lysholm scores, as well as IKDC scores. | Weeks 0-3, 4-6, 7-8, 12 and 16-24 after surgery:

CONTACTS AND LOCATIONS:
Overall Officials: William S Kimmerly, MD, Principal Investigator — Emory University
Locations (1):
- Grady Healthcare System, Atlanta, Georgia, United States